CLINICAL TRIAL: NCT03430830
Title: A Randomized, Open, Three-dose (100 mg, 200 mg and 300 mg) Duplicate Bifunctional Crossover and Fixed 200mg Continuous Dose Study to Evaluate the Pharmacokinetics and Safety of ASC16 Tablets in Healthy Volunteers
Brief Title: A Study to Evaluate the Pharmacokinetics and Safety of ASC16 Tablets in Healthy Volunteers in China
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ascletis Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ASC-ASC16-I-CTP-03
Record Dates: First submitted 2018-01-10; First posted 2018-02-13 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-01

CONDITIONS: Chronic Hepatitis c
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — ravidasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- GROUP 1 (Experimental): 1st day: 2 tablets of Ravidasvir 50mg administered orally once daily; 2nd day: 1 tablet of Ravidasvir 200mg administered orally once daily; 3rd day: 1 tablet of Ravidasvir 200mg and 2 tablets of Ravidasvir 50mg administered orally once daily ; 19th to 25th day： Ravidasvir 200mg administered orally once daily.
  Interventions: Drug: Ravidasvir 50mg; Drug: Ravidasvir 200mg
- GROUP 2 (Experimental): 1st day: Ravidasvir 200mg administered orally once daily; 2nd day: 1 tablet of Ravidasvir 200mg and 2 tablets of Ravidasvir 50mg administered orally once daily ; 3rd day: 2 tablets of Ravidasvir 50mg administered orally once daily; 19th to 25th day：Ravidasvir 200mg administered orally once daily.
  Interventions: Drug: Ravidasvir 50mg; Drug: Ravidasvir 200mg
- GROUP 3 (Experimental): 1st day: 1 tablet of Ravidasvir 200mg and 2 tablets of Ravidasvir 50mg administered orally once daily; 2nd day: 2 tablets of Ravidasvir 50mg administered orally once daily; 3rd day: Ravidasvir 200mg administered orally once daily; 19th to 25th day：Ravidasvir 200mg administered orally once daily.
  Interventions: Drug: Ravidasvir 50mg; Drug: Ravidasvir 200mg
- GROUP 4 (Experimental): 1st day: 1 tablet of Ravidasvir 200mg and 2 tablets of Ravidasvir 50mg administered orally once daily; 2nd day: Ravidasvir 200mg administered orally once daily; 3rd day: 2 tablets of Ravidasvir 50mg administered orally once daily; 19th to 25th day：Ravidasvir 200mg administered orally once daily.
  Interventions: Drug: Ravidasvir 50mg; Drug: Ravidasvir 200mg
- GROUP 5 (Experimental): 1st day: Ravidasvir 200mg administered orally once daily; 2nd day: 2 tablets of Ravidasvir 50mg administered orally once daily; 3rd day: 1 tablet of Ravidasvir 200mg and 2 tablets of Ravidasvir 50mg administered orally once daily; 19th to 25th day：Ravidasvir 200mg administered orally once daily.
  Interventions: Drug: Ravidasvir 50mg; Drug: Ravidasvir 200mg
- GROUP 6 (Experimental): 1st day: 2 tablets of Ravidasvir 50mg administered orally once daily; 2nd day: 1 tablet of Ravidasvir 200mg and 2 tablets of Ravidasvir 50mg administered orally once daily; 3rd day: Ravidasvir 200mg administered orally once daily; 19th to 25th day：Ravidasvir 200mg administered orally once daily.
  Interventions: Drug: Ravidasvir 50mg; Drug: Ravidasvir 200mg

INTERVENTIONS:
Drug: Ravidasvir 50mg — 50mg, Tablet
  Other Names: ASC16
Drug: Ravidasvir 200mg — 200mg, Tablet
  Other Names: ASC16

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics and safety of ASC16 after 3-single dose(50mg、100mg、200mg) or fixed continuous dose(200mg) in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-45 years old;
* Male body weight not less than 50kg; Female body weight not less than 45kg; BMI in the range of 19~24kg/m2
* Healthy men or women based on history, physical examination, laboratory examination and ECG.
* no plan of pregnancy in at least six months, and willing to take effective measures to prevent contraception from the first time when the drug is administered till the last time the drug is administered within 30 days.
* Female has negative pregnancy tests at the screening stage.
* Voluntary to sign the informed consent.

Exclusion Criteria:

* Have medical history, or has disease, such as cardiovascular system, respiratory system, endocrine and metabolic system, urinary system, digestive system, blood system, nerve system disease or psychiatric disease and acute or chronic infectious diseases and malignant tumors.
* Has a history of drug or food allergy.
* Positive hepatitis A antibody，positive hepatitis B surface antigen， positive hepatitis C antibody，syphilis antibody or HIV antibody at screening.
* Laboratory tests out of normal range and judged by the investigators as clinically significant.
* Had gastrointestinal surgery, vagotomy, intestinal resection or any possible interference with gastrointestinal peristalsis, pH or absorbed by surgery.
* Pregnant, lactating women and people who unwilling to take effective measures to prevent contraception.
* People who consumed pomelo, apple or orange and foods or drinks containing their extracted ingredients within 3 days of taking the drug.
* Any prescription or over-the-counter medications, herbs, and vitamins are required to be taken prior to or within the first month of taking the drug.
* Selected within the first 6 months of smoking, alcohol, drug abuse or history of drug abuse.
* Selected within the first 3 months had blood loss or blood donation of 200ml.
* Participate in other clinical trials within the first 3 months of the study and received other study drug treatment.
* In addition to the above, the investigators judged not suitable for participating in this clinical trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2018-04-09 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) | 27 days
  Pharmacokinetics (blood draws, pre- and post-dose)
Area under the plasma concentration versus time curve (AUC) | 27 days
  Pharmacokinetics (blood draws, pre- and post-dose)

CONTACTS AND LOCATIONS:
Overall Officials: Yahong Chen, Master, Study Director — Ascletis Pharmaceuticals Co., Ltd.
Locations (1):
- First Hospital of Zhejiang Province, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu G, Zhou H, Wu J, Lv D, Wu L, Zhai Y, Lin M, Wu JJ, Shentu J. Pharmacokinetics, Safety, and Tolerability of Ravidasvir, with and without Danoprevir/Ritonavir, in Healthy Subjects. Antimicrob Agents Chemother. 2021 Sep 17;65(10):e0060021. doi: 10.1128/AAC.00600-21. Epub 2021 Jul 12. PMID 34252301